CLINICAL TRIAL: NCT00070200
Title: A Pilot Induction Regimen Incorporating Topotecan for Treatment of Newly Diagnosed High Risk Neuroblastoma
Brief Title: Induction Chemotherapy Using Cyclophosphamide and Topotecan in Treating Patients Who Are Undergoing Autologous Peripheral Stem Cell Transplantation for Newly Diagnosed or Progressive Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANBL02P1; CDR0000330140 (Other: Clinical Trials.gov); COG-ANBL02P1 (Other: Children's Oncology Group)
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-02

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma; stage 4S neuroblastoma; localized unresectable neuroblastoma; localized resectable neuroblastoma; regional neuroblastoma; disseminated neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Filgrastim; Cisplatin; Cyclophosphamide; Doxorubicin; Etoposide; Isotretinoin; Melphalan; Topotecan; Vincristine; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): Induction Cycles 1 and 2 (CT) (21 days each), Cyclophosphamide (Days 1 thru 5) weight based dosage (> 12 kg 400 mg/m2/day, < 12 kg 13.3 mg/kg/day, < 2 years old N/A. Topotecan (Days 1 thru 5) weight based dosage (> 12 kg 1.2 mg/m2/day, < 12 kg 0.04 mg/kg/day, < 2 years old 0.04 mg/kg/day). Filgrastim (Days 6 →) weight based dosage (> 12 kg 5 micrograms/kg, < 12 kg 5 micrograms /kg, < 2 years old 5 micrograms /kg.
  Interventions: Biological: filgrastim; Drug: cisplatin; Drug: cyclophosphamide; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: isotretinoin; Drug: melphalan; Drug: topotecan hydrochloride; Drug: vincristine sulfate; Procedure: conventional surgery; Procedure: peripheral blood stem cell transplantation; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim
Drug: cisplatin
Drug: cyclophosphamide
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: isotretinoin
Drug: melphalan
Drug: topotecan hydrochloride
Drug: vincristine sulfate
Procedure: conventional surgery
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as topotecan and cyclophosphamide, use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with autologous stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects of induction chemotherapy using cyclophosphamide and topotecan in treating patients who are undergoing surgery and autologous stem cell transplantation followed by radiation therapy for newly diagnosed or progressive neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the toxicity and feasibility of adding cyclophosphamide and topotecan to induction therapy in patients with newly diagnosed or progressive high-risk neuroblastoma undergoing autologous peripheral blood stem cell (PBSC) transplantation.
* Determine the feasibility of PBSC mobilization and in vivo PBSC tumor purging in these patients after treatment with this regimen.

Secondary

* Determine tumor response rate in patients treated with this regimen.
* Determine the pharmacokinetics of this regimen in these patients.
* Determine whether topotecan affects cyclophosphamide pharmacokinetics in these patients.
* Correlate host DNA with toxicity and cyclophosphamide and topotecan pharmacokinetics in patients treated with this regimen.
* Determine toxicity in patients treated with this regimen.

OUTLINE: This is a pilot, multicenter study. Patients are stratified according to diagnosis (newly diagnosed vs initially stage 1, 2, or 4S that progressed to stage 4 without interval chemotherapy).

* Induction therapy: Patients receive 6 courses of induction therapy.

  * Courses 1 and 2: Patients receive cyclophosphamide IV over 30 minutes and topotecan IV over 30 minutes on days 1-5 and filgrastim (G-CSF) subcutaneously (SC) or IV beginning on day 6 and continuing until blood counts recover.
  * Course 3: Patients receive etoposide IV over 2 hours on days 1-3, cisplatin IV over 1 hour on days 1-4, and G-CSF SC or IV beginning on day 5 and continuing until blood counts recover.
  * Course 4: Patients receive cyclophosphamide IV over 6 hours on day 1 and doxorubicin IV and vincristine IV continuously over 24 hours on days 1-3. Patients also receive G-CSF SC or IV beginning on day 4 and continuing until blood counts recover.
  * Course 5: Patients receive etoposide, cisplatin, and G-CSF as in course 3.
  * Course 6: Patients receive cyclophosphamide, doxorubicin, vincristine, and G-CSF as in course 4.

Treatment repeats every 21 days for a total of 6 courses in the absence of disease progression or unacceptable toxicity.

* Consolidation therapy: Within 4-6 weeks after completing induction therapy, patients receive melphalan IV on days -7 to -5 and etoposide IV and carboplatin IV continuously over 24 hours on days -7 to -4.
* Stem cell transplantation: Peripheral blood stem cells are collected after course 2 of induction therapy and infused on day 0. Patients receive G-CSF IV beginning on day 0 and continuing until blood counts recover.
* Surgery: After course 5 of induction therapy, patients undergo surgery.
* Radiotherapy: Beginning 28-42 days after transplantation, patients receive 12 fractions of local radiotherapy to all areas of residual soft tissue disease and the primary tumor site, even if completely resected.
* Maintenance therapy: Beginning 66 days after transplantation, patients receive oral isotretinoin twice daily on days 1-14. Treatment repeats every 28 days for a total of 6 courses.

Patients are followed every 3 months for 1 year, every 6 months for 4 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 10-29 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed neuroblastoma or ganglioneuroblastoma meeting 1 of the following staging criteria:

  * Newly diagnosed disease, at least 1 year of age, and meets criteria for 1 of the following:

    * International Neuroblastoma Staging System (INSS) stage 2a/2b with MYCN amplification (greater than 10) AND unfavorable pathology
    * INSS stage 3 with MYCN amplification OR unfavorable pathology
  * Newly diagnosed INSS stage 4 disease meeting criteria for 1 of the following:

    * Over 18 months of age
    * Age 12 to 18 months with any unfavorable biologic feature (MYCN amplification, unfavorable pathology, and/or DNA index=1) or any biologic feature that is indeterminant, unsatisfactory, or unknown

      * No INSS stage 4 disease and age 12 to 18 months with all 3 favorable biologic features (i.e., nonamplified MYCN, favorable pathology, and DNA index greater than 1)
  * Newly diagnosed INSS stage 3, 4, or 4S disease AND under 1 year of age with MYCN amplification
  * At least 1 year of age and initially diagnosed with INSS stage 1, 2, or 4S disease that progressed to stage 4 without interval chemotherapy

    * Must have been enrolled on COG-ANBL00B1 at initial diagnosis

PATIENT CHARACTERISTICS:

Age

* 30 and under at initial diagnosis

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count at least 1,000/mm^3*
* Platelet count at least 100,000/mm^3* (transfusion independent)
* Hemoglobin at least 10.0 g/dL* (red blood cell transfusions allowed) NOTE: *Granulocytopenia, anemia, and/or thrombocytopenia allowed for patients with tumor metastatic to the bone marrow

Hepatic

* Bilirubin no greater than 1.5 mg/dL
* ALT less than 300 IU/L

Renal

* Creatinine no greater than 1.5 mg/dL
* Creatinine clearance or radioisotope glomerular filtration rate at least 60 mL/min

Cardiovascular

* ECG normal
* Shortening fraction at least 27% by echocardiogram OR
* Ejection fraction at least 50% by MUGA

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* See Disease Characteristics
* No more than 1 prior chemotherapy course on the low- or intermediate-risk neuroblastoma studies (COG-P9641, COG-A3961) prior to determination of MYCN amplification and Shimada histology

Endocrine therapy

* Not specified

Radiotherapy

* Prior localized emergency radiotherapy to sites of life-threatening or function-threatening disease allowed

Surgery

* Not specified

Other

* No other prior systemic therapy

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2004-03; Primary Completion 2006-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are classified as a "success" | Length of study
  Given that the documented delivered dose intensity of chemotherapy in current induction regimens is 75-85% of the intended dose intensity,5,78 we shall consider an individual patient as a "success" in terms of feasibility if the patient is able to receive 75% or more of the intended chemotherapy doses of known active agents.

SECONDARY OUTCOMES:
Number of toxic deaths | Length of study
Proportion of patients with dose limiting toxicities during induction cycle 1 and 2 | Length of study
  Dose limiting toxicities during induction cycle 1 and 2 will be used to modify the topotecan dosage if necessary and to address Primary Aim 1 in a descriptive fashion.
Tumor contamination of PBSCs | Length of study
  Tumor contamination of PBSCs as measured by immunohistochemical analysis following cycle 2 induction;
Inability to adequately mobilize PBSCs | Length of study
  Inability to adequately mobilize PBSCs, defined as a harvest of < 1.5 x 10 6 CD 34 cells/kg. A patient will be designated a PBSCs "failure" if either a) or b) is the case.
Assessment of response | Length of study
  After completion of induction therapy. Response will be determined using the International Response Criteria defined elsewhere in the protocol. The tumor response rate will be defined as the proportion of patients who achieve a CR, VGPR, or PR after completion of induction therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Julie R. Park, MD, Study Chair — Seattle Children's Hospital
Locations (6):
- United States (5):
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Children's Hospital and Regional Medical Center - Seattle, Seattle, Washington
  - Mary Bridge Children's Hospital and Health Center - Tacoma, Tacoma, Washington
- Westmead Hospital, Westmead, New South Wales, Australia

REFERENCES:
- [Result] Park JR, Scott JR, Stewart CF, London WB, Naranjo A, Santana VM, Shaw PJ, Cohn SL, Matthay KK. Pilot induction regimen incorporating pharmacokinetically guided topotecan for treatment of newly diagnosed high-risk neuroblastoma: a Children's Oncology Group study. J Clin Oncol. 2011 Nov 20;29(33):4351-7. doi: 10.1200/JCO.2010.34.3293. Epub 2011 Oct 17. PMID 22010014